CLINICAL TRIAL: NCT03551873
Title: A Phase 4 Open-label, Non-randomized Study Evaluating the Pharmacokinetics and Safety of TRULANCE® (Plecanatide) in Breast Milk of Lactating Women Treated With TRULANCE
Brief Title: A Postmarketing Study of Plecanatide in Breast Milk of Lactating Women Treated With TRULANCE®
Status: Completed | Type: Observational
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: SP304-3117-14
Record Dates: First submitted 2018-04-19; First posted 2018-06-11 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Chronic Idiopathic Constipation
Keywords: Breast milk; Lactating
MeSH Terms: interventions — plecanatide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Breast milk
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes

INTERVENTIONS:
Drug: Plecanatide — Subjects will have been breastfeeding or pumping for at least 4 weeks and must have been prescribed and taking TRULANCE® for at least 14 continuous days prior to Baseline. Breast milk for measurement of TRULANCE® (plecanatide) concentrations will be collected at Day 1.
  Other Names: TRULANCE®

SUMMARY:
This is a multi-center, open-label study evaluating pharmacokinetics of TRULANCE® (plecanatide) in breast milk of lactating women treated with TRULANCE

DETAILED DESCRIPTION:
This is an open-label study in lactating women who have been prescribed TRULANCE® by their healthcare provider. The study will assess the pharmacokinetics of plecanatide and its active metabolite in breast milk of lactating women treated therapeutically with TRULANCE. Subjects will be screened prior to admission for Baseline assessments. Following final qualifications, the morning dose of TRULANCE will be administered under supervision from study personnel and serial samples of breast milk will be collected via breast pump.

ELIGIBILITY:
Inclusion Criteria:

* Females ≥ 18 years of age
* Has been breastfeeding or actively pumping for at least 4 weeks
* Has been prescribed TRULANCE by a healthcare provider and has taken it for a minimum of 14 consecutive days before anticipated Baseline Visit
* Has the ability to understand and communicate the requirements of the study and is willing to continue breastfeeding or regular pumping in order to maintain milk supply for the duration of the study
* Weaning must not be underway

Exclusion Criteria:

* Has clinically significant medical or psychiatric condition (as determined by the Medical Monitor) other than the medical condition being treated with TRULANCE
* Has mastitis or other condition that would prevent the collection of milk from one or both breasts.
* Has participated in an investigational drug study within the 90 days prior to CRU admission

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Lactating women with Chronic idiopathic Constipation (CIC) or Irritable Bowel Syndrome with Constipation (IBS-C)
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2018-12-14 (Actual); Study Completion 2018-12-14 (Actual)

PRIMARY OUTCOMES:
Cmax,ss of TRULANCE (plecanatid) and its active metabolite in breast milk | Day 1 (pre-dose [1 hour before dosing], at 2, 6 and 12 hours post-dose)
  Maximum observed concentration of TRULANCE (plecanatide) in breast milk during a dosing interval at steady state
Cavg,ss of TRULANCE (plecanatide) and its active metabolite in breast milk | Day 1 (pre-dose [1 hour before dosing], at 2, 6 and 12 hours post-dose)
  Average concentration of TRULANCE (plecanatide) in breast milk at steady state
AUCτ,ss of TRULANCE (plecanatide) and its active metabolite in breast milk | Day 1 (pre-dose [1 hour before dosing], at 2, 6 and 12 hours post-dose)
  Area under the concentration-time curve during a dosing interval at steady state interval at steady state
Aτ,ss of TRULANCE (plecanatide) and its active metabolite in breast milk | Day 1 (pre-dose [1 hour before dosing], at 2, 6 and 12 hours post-dose)
  Amount (of unchanged drug) excreted into the milk during a dosing interval at steady state a dosing interval (τ) at steady state

CONTACTS AND LOCATIONS:
Overall Officials: Anhthu Nguyen, Study Director — Synergy Pharmaceuticals Inc.
Locations (3):
- United States (3):
  - Synergy Research Center 002, North Hollywood, California
  - Syergy Research Center 003, Tamarac, Florida
  - Synergy Research Center 001, Raleigh, North Carolina